CLINICAL TRIAL: NCT01677455
Title: An Open-Label Multicenter Phase 2 Window of Opportunity Study Evaluating Ganetespib in Women With Breast Cancer
Acronym: Enchant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9090-11
Record Dates: First submitted 2012-07-09; First posted 2012-09-03 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer; HER-2 Positive Breast Cancer; Triple Negative Breast Cancer; ER/Progressive Response (PR) + Refractory to Prior Hormonal Treatment
Keywords: Hsp90 inhibitor; ganetespib; STA 9090
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HER2+ breast cancer (Experimental)
  Interventions: Drug: ganetespib
- Triple negative breast cancer (Experimental): Closed to enrollment
  Interventions: Drug: ganetespib
- ER/PR+ Refractory to Prior Hormonal Treatment (Experimental)
  Interventions: Drug: ganetespib

INTERVENTIONS:
Drug: ganetespib — Ganetespib 150 mg/m2 will be administered intravenously, twice weekly, for three consecutive weeks of each 4 week cycle.

SUMMARY:
The purpose of this study is to determine if ganetespib (STA-9090) is effective in the treatment of patients with HER2+ or triple negative breast cancer who have not received prior systemic treatment in the metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of invasive breast cancer.
* Stage IV disease.
* Documented HER2 and hormonal receptor status per protocol, ER/PR+ patients must be refractory to at least one prior hormonal treatment.
* ECOG Performance status 0-1.
* Measurable disease per RECIST (1.1).
* Adequate hematological function per protocol.
* Adequate hepatic function per protocol.
* Adequate renal function per protocol.
* Negative serum pregnancy test at study entry for patients of childbearing potential.
* Ability to understand and sign written consent and to comply with the study protocol.

Exclusion Criteria:

* Presence of active or untreated CNS metastases as determined by MRI/CT scan performed during screening.
* Active malignancies other than MBC within the last 5 years except adequately treated in situ carcinoma of the cervix uteri or basal or squamous cell carcinoma of the skin.
* Bone as the only site of metastatic disease from breast cancer.
* Prior radiotherapy to the only area of measurable disease. NOTE: Radiotherapy to a limited area other than the sole site of measurable disease is allowed, if received prior to initiation of ganetespib treatment. Patients must have completed treatment and recovered from all acute treatment-related toxicities prior to administration of first dose of ganetespib.
* Pregnancy or lactation.
* Known serious cardiac illness.
* Uncontrolled intercurrent illness per protocol.
* Other severe acute or chronic medical condition or abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, or that in the judgment of the investigator would make the patient inappropriate for entry into the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-07; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Week 12
  Objective response rate is based on RECIST criteria

SECONDARY OUTCOMES:
Duration of response and progression free survival | Every six weeks until progression
  Progressive disease based on RECIST criteria. CT scans at week 6, week 12 and every 6 weeks thereafter for the duration of the study.

CONTACTS AND LOCATIONS:
Locations (25):
- United States (8):
  - Synta Pharmaceuticals Investigative Site, Birmingham, Alabama
  - Synta Pharmaceuticals Investigative Site, Altanta, Georgia
  - Synta Pharmaceuticals Investigative Site, Boston, Massachusetts
  - Synta Pharmaceuticals Investigative Site, New York, New York
  - Synta Pharmaceuticals Investigative Site, Durham, North Carolina
  - Synta Pharmaceuticals Investigative Site, Columbus, Ohio
  - Synta Pharmaceuticals Investigative Site, Philadelphia, Pennsylvania
  - Synta Pharmaceutical Investigative Site, Houston, Texas
- Argentina (2):
  - Synta Pharmaceuticals Investigative Site, Córdoba
  - Synta Pharmaceuticals Investigative Site, Rosario Santa Fe
- Belgium (3):
  - Synta Pharmaceuticals Investigative Site, Brussels
  - Synta Pharmaceutical Investigative Site, Charleroi
  - Synta Pharmaceuticals Investigative Site, Wilrijk
- Synta Pharmaceuticals Investigative Site, São Paulo, Brazil
- Synta Pharmaceuticals Investigative Site, Lima, Peru
- South Korea (4):
  - Synta Pharmaceutical Investigative Site, Seoul, Gangnam-GU
  - Synta Pharmaceuticals Investigative Site, Seoul, Jongno-Gu
  - Synta Pharmacuetical Investigative Site, Seoul, Seodaemun-GU
  - Synta Pharmaceuticals Investigative Site, Seoul, Songpa-Gu
- Synta Pharmaceuticals Investigative Site, Barcelona, Spain
- United Kingdom (5):
  - Synta Pharmaceutical Investigative Site, Edinburgh
  - Synta Pharmaceutical Investigative Site, Glasgow
  - Synta Pharmaceutical Investigative Site, Nottingham
  - Synta Pharmaceuticals Investigative Site, Oxford
  - Synta Pharmaceutical Investigative Site, Peterborough